CLINICAL TRIAL: NCT01178190
Title: The Diagnostic Yield of Narrow Band Imaging Videobronchoscopy in Lung Cancer
Brief Title: The Role of Narrow Band Imaging Videobronchoscopy in Lung Cancer
Acronym: NBI
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Chang Min ,Choi, Asan medical center
Other Study IDs: NBI-AMC
Record Dates: First submitted 2010-07-28; First posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-06

CONDITIONS: Lung Cancer
Keywords: narrow band imaging; malignant lesion; lung cancer; NBI
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- lung cancer

SUMMARY:
Narrow band imaging (NBI) videobronchoscopy is an optical technique in which filtered light enhances superficial neoplasm based on their neoangiogenic pattern. The objectives of this study investigate its better diagnostic yield in the assessment of lung cancer than conventional flexible bronchoscopy.

DETAILED DESCRIPTION:
Inspection with high resolution endoscopy was followed by NBI. Detected lesions were biopsied. applied the system of shibuya et al. to analyze and classify vascular patterns by NBI into four categories (spiral and screw pattern, dotted pattern, tortuous pattern, avascular pattern) compared with the known diagnostic yield of conventional white light bronchoscopy, An equivalent or superior result will also significantly impact on patient care This technology could aid not only early-stage lung cancer diagnosis but also more accurate local staging of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* endobronchial lesion on chest CT

Exclusion Criteria:

* Age < 18 years old
* Inability to consent for the study
* Inability to tolerate bronchoscopy
* Active pulmonary infection (bronchitis, pneumonia)
* ST elevation or depression on ECG
* Prothrombin time prolongation(<70%)
* platelet <10,000

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: suspected endobroncheal lesion on chest CT
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
accuracy of NBI videobronchoscopic biopsy | 10-11 months
  Define and compare the sensitivity, specificity, positive predictive value, negative predictive value, likelihood ratio and accuriacies for the diagnostic techniques for lung cancer.

SECONDARY OUTCOMES:
early cancer lesion detection rate using Shibuya descriptors | 10-11 months
  Define and compare the sensitivity, specificity, positive predictive value, negative predictive value, likelihood ratio and accuriacies for the diagnostic techniques for early lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: ChangMin Choi, M.D., Principal Investigator — Asan Medical Center
Locations (1):
- ChangMin, Choi, Seoul, Seoul, South Korea